CLINICAL TRIAL: NCT04074876
Title: Utility of Pulmonary Echography for Evaluation of Patients Undergoing Orthopedic Surgery for Femur Fracture
Acronym: LUSHIP
Status: Completed | Type: Observational
Sponsor: University of Udine (Other)
Responsible Party: Principal Investigator, Tiziana Bove, Professor, University of Udine
Other Study IDs: Lung US orthopedic surgery
Record Dates: First submitted 2019-08-12; First posted 2019-08-30 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Femur Fracture
Keywords: pulmonary ultrasound; urgency orthopedic surgery; major adverse cardiac events
MeSH Terms: conditions — Femoral Fractures; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with femur fracture: Group is composed of patients more of 65 years of age with femur fracture undergoing urgent orthopedic surgery.
  During normal pre-operative evaluation and classification based on principal scores and laboratory data, patients will be subjected to bedside pulmonary ultrasound.
  Pulmonary ultrasound will evaluate the presence of one of four patterns (normal pattern, isolated B lines, coalescent B lines and consolidation) defined by Lung Ultrasound Score in the 6 fields for each hemithorax of the patient.
  These patients will be later subjected to spinal anaesthesia and orthopedic surgery.
  They will be follow for evaluation of MACE (major adverse cardiovascular events: atrial fibrillation, flutter, acute heart failure and non-fatal acute myocardial infarction)
  Interventions: Device: Pulmonary echography

INTERVENTIONS:
Device: Pulmonary echography — Pulmonary echography during preoperative evaluation for patients undergoing urgency orthopedic surgery for femur fracture.
  Pulmonary ultrasound will evaluate the presence of one of four patterns defined by Lung Ultrasound Score in the 6 fields for each hemithorax of the patient (2 anterior, 2 lateral and 2 posterior). Each region is defined by axillary lines (anterior and posterior) and then is divided into 2 subregions (superior and inferior), thus defining the 6 fields. For a comprehensive exam, all intercostal spaces in the setting of each field will have to be examined by sliding the probe along them . A score will be used for each field that will have this definition:
  * 0: normal pattern (A-lines)
  * 1: multiple B lines (at least 3 for field), well defined.
  * 2: B lines coalescent
  * 3: consolidation of any dimension

SUMMARY:
The stratification of perioperative risk is an essential moment in the preoperative evaluation of the patient undergoing surgery especially in the setting of urgency. There is a very broad group of indexes used in the stratification of preoperative risk, like ASA-PS (American Society of Anesthesiologists Physical Status), RCRI (Revised Cardiac Risk Index) and NSQIP MICA (National Surgical Quality Improvement Program Myocardial Infarction or Cardiac Arrest). The role of some laboratory markers such as BNP has also been demonstrated. The fundamental point of all these scores is cardiocirculatory compensation.

There are concerns about the value of certain preoperative exams, especially in an urgent setting. Of them all, mostly chest X-ray is questioned. Chest X-ray, indeed, needs special costs, not always short execution times and the need for X-ray exposition. Furthermore, its utility is questionable in asymptomatic patients, in which there are often no alterations to be detected. Sensibility, for Thorax x-ray, is 41% for apical flow inversion, 27% for interstitial and 6% for alveolar oedema. In chronic decompensated patients, radiographic signs of congestion have a small diagnostic accuracy, being absent in 53% of patients with capillary pulmonary pressure between 16 and 29 mmHg and in 39% of those with wedge pressure more of 30 mmHg.

Pulmonary echography is a known method, that has different possible applications in diagnosis of the lung parenchymal and pleural disease.

Lung is made up for 80% of water. Extravascular lung water is physiologically less than 500 ml and it increases in the case of pathology. Augmentation of this water is detected reliably by echography.

B-lines are an echographic artefact that allows recognition of interstitial syndrome, having a sensibility of 93,4% and specificity of 93%. Presence of 3 or more of B-lines in 2 out of 4 fields of each hemithorax can identify a cardiac problem like pulmonary sub-oedema or chronic heart failure and it is known as Diffuse Interstitial Syndrome. Thorax X-ray, instead, detects these situations only when extravascular water exceeds 30%. That's why echography has been proposed as a method for evaluation of extravascular pulmonary water. Moreover, when lung air component is lost enough in subpleural area, it is possible to find little consolidations. A method of reporting different grades of loss of aeration of the lung (normal pattern, isolated B lines, coalescent B lines and consolidation) has been proposed as a tool for monitoring the aeration itself.

Pleural effusion is another sign that echography could detect. It is perfectly transonic and easy to see. Also, in this case, therefore, ultrasound is superior to X-ray, that has got sensibility, specificity and diagnostic accuracy of 67%, 70% and 67% respectively.

All this information could provide useful elements for preoperative patient management. Echography, indeed, is a bedside and real-time method, that can give rapid information about the cardiocirculatory situation of patients.

Using this method, that is non-invasive and easy, useful elements could be obtained, that could contribute to a better overview of clinical conditions of the patient in the preoperative setting.

In the particular field of urgency and, among all, in the setting of orthopaedic urgency for femur fracture, there is a need for a more rapid and comprehensive evaluation, giving that the patient has to be operated within 24-48 hours. This timing is often incompatible with a long and time-consuming evaluation of the patients. Furthermore, a complete cardiologic examination is beyond the requirements of international guidelines for intermediate surgery, since it doesn't change the perioperative management.

In this particular setting, hence, pulmonary echography could represent a more reliable and easier tool compared to thorax X-ray, often performed in non-optimal conditions (supine position, only anteroposterior chest X-ray).

In recent studies, percentage of major adverse cardiovascular events (atrial fibrillation, flutter, acute heart failure and non-fatal acute myocardial infarction) after hip fracture has settled around 24.8%. This data confirms the importance of a valid preoperative stratification in this setting.

From this perspective, this study aims to evaluate the utility of pulmonary echography as a preoperative method of investigation.

The principal aim is to evaluate the utility of the pulmonary echography in predicting the risk of patients undergoing urgent surgery for femur fracture.

Alternative objectives are:

* Evaluate the predictability of LUS (lung ultrasound score) on the occurrence of MACE (major adverse cardiovascular events)
* Verify feasibility of echographic evaluation in the estimation of fluid tolerance of patients undergoing orthopaedic surgery.
* Evaluation of postoperative pulmonary complications (PPC)

ELIGIBILITY:
Inclusion Criteria:

* Patients more of 65 years of age with femur fracture undergoing urgent surgery
* patients can undergo spinal anaesthesia

Exclusion Criteria:

* Absent consent, patients with acute heart failure or recent major cardiac events (< 6 months), known pulmonary parenchyma diseases (including pneumonia), general anaesthesia during surgery

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study will be conducted between the patients hospitalized in the Orthopaedic Ward of Udine's Hospital and other participating centres, because of femur fracture undergoing urgent surgery. Anesthesiology management will be in charge of the physicians of Anesthesiology Division of the same Hospital, according to the international guidelines concerning preoperative evaluation.
Sampling Method: Non-Probability Sample
Enrollment: 877 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2022-09-21 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Accuracy of ultrasound in predicting MACE (major adverse cardiovascular events) in the setting of the study | pulmonary echography is made during pre-operative anesthesiologic evaluation, patients are in follow up for MACE for 30 days
  Patients are classified by echography pattern in four category (normal pattern (A-lines), well defined multiple B lines (at least 3 for field), B lines coalescent, consolidation of any dimension). After surgery, the occurrence of MACE during the whole follow-up period will be evaluate in the four category of patients.

SECONDARY OUTCOMES:
Feasibility of echography in evaluation of the tolerance to fluid challenge during surgery | pulmonary echography is made during pre-operative anesthesiologic evaluation, patients are evaluated during surgery for fluid tollerance
  Estimate a correlation between echography and fluid challenge during surgery
finding postoperative pulmonary complications | pulmonary echography is made during pre-operative anesthesiologic evaluation, patients are in follow up for postoperative pulmonary complications for 30 days
  Follow up for patients after orthopedic surgery and value consecutive pulmonary complications

CONTACTS AND LOCATIONS:
Locations (1):
- S. Maria della Misericordia Hospital, Udine, Italy

REFERENCES:
- [Background] Hendrix JM, Garmon EH. American Society of Anesthesiologists Physical Status Classification System. 2025 Feb 11. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK441940/ PMID 28722969
- [Background] Lee TH, Marcantonio ER, Mangione CM, Thomas EJ, Polanczyk CA, Cook EF, Sugarbaker DJ, Donaldson MC, Poss R, Ho KK, Ludwig LE, Pedan A, Goldman L. Derivation and prospective validation of a simple index for prediction of cardiac risk of major noncardiac surgery. Circulation. 1999 Sep 7;100(10):1043-9. doi: 10.1161/01.cir.100.10.1043. PMID 10477528
- [Background] Fleisher LA, Beckman JA, Brown KA, Calkins H, Chaikof EL, Fleischmann KE, Freeman WK, Froehlich JB, Kasper EK, Kersten JR, Riegel B, Robb JF, Smith SC Jr, Jacobs AK, Adams CD, Anderson JL, Antman EM, Buller CE, Creager MA, Ettinger SM, Faxon DP, Fuster V, Halperin JL, Hiratzka LF, Hunt SA, Lytle BW, Nishimura R, Ornato JP, Page RL, Riegel B, Tarkington LG, Yancy CW. ACC/AHA 2007 Guidelines on Perioperative Cardiovascular Evaluation and Care for Noncardiac Surgery: Executive Summary: A Report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Writing Committee to Revise the 2002 Guidelines on Perioperative Cardiovascular Evaluation for Noncardiac Surgery) Developed in Collaboration With the American Society of Echocardiography, American Society of Nuclear Cardiology, Heart Rhythm Society, Society of Cardiovascular Anesthesiologists, Society for Cardiovascular Angiography and Interventions, Society for Vascular Medicine and Biology, and Society for Vascular Surgery. J Am Coll Cardiol. 2007 Oct 23;50(17):1707-32. doi: 10.1016/j.jacc.2007.09.001. No abstract available. PMID 17950159
- [Background] Gupta PK, Gupta H, Sundaram A, Kaushik M, Fang X, Miller WJ, Esterbrooks DJ, Hunter CB, Pipinos II, Johanning JM, Lynch TG, Forse RA, Mohiuddin SM, Mooss AN. Development and validation of a risk calculator for prediction of cardiac risk after surgery. Circulation. 2011 Jul 26;124(4):381-7. doi: 10.1161/CIRCULATIONAHA.110.015701. Epub 2011 Jul 5. PMID 21730309
- [Background] De Hert S, Staender S, Fritsch G, Hinkelbein J, Afshari A, Bettelli G, Bock M, Chew MS, Coburn M, De Robertis E, Drinhaus H, Feldheiser A, Geldner G, Lahner D, Macas A, Neuhaus C, Rauch S, Santos-Ampuero MA, Solca M, Tanha N, Traskaite V, Wagner G, Wappler F. Pre-operative evaluation of adults undergoing elective noncardiac surgery: Updated guideline from the European Society of Anaesthesiology. Eur J Anaesthesiol. 2018 Jun;35(6):407-465. doi: 10.1097/EJA.0000000000000817. PMID 29708905
- [Background] Vetrugno L, Langiano N, Gisonni R, Rizzardo A, Venchiarutti PE, Divella M, Pompei L, Causero A, Rocca GD. Prediction of early postoperative major cardiac events after elective orthopedic surgery: the role of B-type natriuretic peptide, the revised cardiac risk index, and ASA class. BMC Anesthesiol. 2014 Mar 21;14:20. doi: 10.1186/1471-2253-14-20. PMID 24655733
- [Background] O'Neill F, Carter E, Pink N, Smith I. Routine preoperative tests for elective surgery: summary of updated NICE guidance. BMJ. 2016 Jul 14;354:i3292. doi: 10.1136/bmj.i3292. No abstract available. PMID 27418436
- [Background] Knudsen CW, Omland T, Clopton P, Westheim A, Abraham WT, Storrow AB, McCord J, Nowak RM, Aumont MC, Duc P, Hollander JE, Wu AH, McCullough PA, Maisel AS. Diagnostic value of B-Type natriuretic peptide and chest radiographic findings in patients with acute dyspnea. Am J Med. 2004 Mar 15;116(6):363-8. doi: 10.1016/j.amjmed.2003.10.028. PMID 15006584
- [Background] Chakko S, Woska D, Martinez H, de Marchena E, Futterman L, Kessler KM, Myerberg RJ. Clinical, radiographic, and hemodynamic correlations in chronic congestive heart failure: conflicting results may lead to inappropriate care. Am J Med. 1991 Mar;90(3):353-9. doi: 10.1016/0002-9343(91)80016-f. PMID 1825901
- [Background] Lichtenstein DA. Lung ultrasound in the critically ill. Ann Intensive Care. 2014 Jan 9;4(1):1. doi: 10.1186/2110-5820-4-1. PMID 24401163
- [Background] Volpicelli G, Elbarbary M, Blaivas M, Lichtenstein DA, Mathis G, Kirkpatrick AW, Melniker L, Gargani L, Noble VE, Via G, Dean A, Tsung JW, Soldati G, Copetti R, Bouhemad B, Reissig A, Agricola E, Rouby JJ, Arbelot C, Liteplo A, Sargsyan A, Silva F, Hoppmann R, Breitkreutz R, Seibel A, Neri L, Storti E, Petrovic T; International Liaison Committee on Lung Ultrasound (ILC-LUS) for International Consensus Conference on Lung Ultrasound (ICC-LUS). International evidence-based recommendations for point-of-care lung ultrasound. Intensive Care Med. 2012 Apr;38(4):577-91. doi: 10.1007/s00134-012-2513-4. Epub 2012 Mar 6. PMID 22392031
- [Background] Agricola E, Picano E, Oppizzi M, Pisani M, Meris A, Fragasso G, Margonato A. Assessment of stress-induced pulmonary interstitial edema by chest ultrasound during exercise echocardiography and its correlation with left ventricular function. J Am Soc Echocardiogr. 2006 Apr;19(4):457-63. doi: 10.1016/j.echo.2005.11.013. PMID 16581487
- [Background] Volpicelli G, Skurzak S, Boero E, Carpinteri G, Tengattini M, Stefanone V, Luberto L, Anile A, Cerutti E, Radeschi G, Frascisco MF. Lung ultrasound predicts well extravascular lung water but is of limited usefulness in the prediction of wedge pressure. Anesthesiology. 2014 Aug;121(2):320-7. doi: 10.1097/ALN.0000000000000300. PMID 24821071
- [Background] Bouhemad B, Brisson H, Le-Guen M, Arbelot C, Lu Q, Rouby JJ. Bedside ultrasound assessment of positive end-expiratory pressure-induced lung recruitment. Am J Respir Crit Care Med. 2011 Feb 1;183(3):341-7. doi: 10.1164/rccm.201003-0369OC. Epub 2010 Sep 17. PMID 20851923
- [Background] Kataoka H. Ultrasound pleural effusion sign as a useful marker for identifying heart failure worsening in established heart failure patients during follow-up. Congest Heart Fail. 2012 Sep-Oct;18(5):272-7. doi: 10.1111/j.1751-7133.2012.00285.x. Epub 2012 Mar 13. PMID 22994441
- [Background] Dogan V, Biteker M, Ozlek E, Ozlek B, Basaran O, Yildirim B, Kayatas K, Celik O, Dogan MM. Impact of preoperative cardiology consultation prior to intermediate-risk surgical procedures. Eur J Clin Invest. 2018 Sep;48(9):e12794. doi: 10.1111/eci.12794. Epub 2018 Jul 25. PMID 28783209
- [Background] Matot I, Oppenheim-Eden A, Ratrot R, Baranova J, Davidson E, Eylon S, Peyser A, Liebergall M. Preoperative cardiac events in elderly patients with hip fracture randomized to epidural or conventional analgesia. Anesthesiology. 2003 Jan;98(1):156-63. doi: 10.1097/00000542-200301000-00025. PMID 12502992
- [Background] Kim BS, Kim TH, Oh JH, Kwon CH, Kim SH, Kim HJ, Hwang HK, Chung SM. Association between preoperative high sensitive troponin I levels and cardiovascular events after hip fracture surgery in the elderly. J Geriatr Cardiol. 2018 Mar;15(3):215-221. doi: 10.11909/j.issn.1671-5411.2018.03.002. PMID 29721000
- [Background] Bouhemad B, Mongodi S, Via G, Rouquette I. Ultrasound for "lung monitoring" of ventilated patients. Anesthesiology. 2015 Feb;122(2):437-47. doi: 10.1097/ALN.0000000000000558. No abstract available. PMID 25501898
- [Derived] Vetrugno L, Boero E, Berchialla P, Forfori F, Bernardinetti M, Spadaro S, Cammarota G, Bruni A, Garofalo E, Tescione M, Deana C, Federici N, Mattuzzi L, Meroi F, Flaibani L, Cortegiani A, Longhini F, Cavarape A, Biasucci DG, D'Inca S, Pesamosca A, Cattarossi A, Granzotti S, D'Orlando L, Urso F, Colombotto C, Tuinman PR, De Robertis E, Livigni S, Maggiore SM, Ranieri VM, Bignami EG; LUSHIP Study Group; Active Ageing interdisciplinary Team. Accuracy of preoperative lung ultrasound score for the prediction of major adverse cardiac events in elderly patients undergoing HIP surgery under spinal anesthesia: The LUSHIP multicenter observational prospective study. Anaesth Crit Care Pain Med. 2024 Dec;43(6):101432. doi: 10.1016/j.accpm.2024.101432. Epub 2024 Oct 5. PMID 39369987
- [Derived] Vetrugno L, Boero E, Bignami E, Cortegiani A, Raineri SM, Spadaro S, Moro F, D'Inca S, D'Orlando L, Agro FE, Bernardinetti M, Forfori F, Corradi F, Pregnolato S, Mosconi M, Bellini V, Franchi F, Mongelli P, Leonardi S, Giuffrida C, Tescione M, Bruni A, Garofalo E, Longhini F, Cammarota G, De Robertis E, Giglio G, Urso F, Bove T; LUSHIP Study Investigators. Association between preoperative evaluation with lung ultrasound and outcome in frail elderly patients undergoing orthopedic surgery for hip fractures: study protocol for an Italian multicenter observational prospective study (LUSHIP). Ultrasound J. 2021 Jun 7;13(1):30. doi: 10.1186/s13089-021-00230-w. PMID 34100124